CLINICAL TRIAL: NCT07305831
Title: A Double-Blind, Placebo-Controlled Trial to Evaluate the Effect of MK-8507 on the QTc Interval in Healthy Adult Participants
Brief Title: A Clinical Trial to Evaluate the Effect of Ulonivirine (MK-8507) on Heart Rhythm in Healthy Adults (MK-8507-012)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 8507-012; MK-8507-012 (Other: MSD)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — ulonivirine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxifloxacin 400 mg + Placebo (Arm 1) (Experimental): Participants will receive ulonivirine dose matched placebo + moxifloxacin dose matched placebo OR ulonivirine dose matched placebo + moxifloxacin 400 mg.
  Interventions: Drug: Moxifloxacin; Drug: Ulonivirine Placebo; Drug: Moxifloxacin Placebo
- Ulonivirine Dose 1 + Placebo (Arm 2) (Experimental): Participants will receive ulonivirine dose matched placebo + moxifloxacin dose matched placebo OR moxifloxacin dose matched placebo + ulonivirine Dose 1.
  Interventions: Drug: Ulonivirine; Drug: Ulonivirine Placebo; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Ulonivirine — Oral tablet
  Other Names: MK-8507; ULO
  Arms: Ulonivirine Dose 1 + Placebo (Arm 2)
Drug: Moxifloxacin — Oral tablet
  Arms: Moxifloxacin 400 mg + Placebo (Arm 1)
Drug: Ulonivirine Placebo — Oral tablet
Drug: Moxifloxacin Placebo — Oral tablet

SUMMARY:
Researchers are looking for new treatments for HIV-1 (human immunodeficiency virus type 1) that are safe, well-tolerated, and can be taken less often. HIV-1 is the most common type of HIV, which is a virus that attacks cells of the immune system.

Ulonivirine (MK-8507) is a study medicine designed to treat HIV-1

The goal of this study is to learn if ulonivirine does not increase the QT interval (a measure of heart rhythm on an electrocardiogram) above a certain amount. Researchers also want to learn what happens to the amount of ulonivirine in a healthy person's body over time.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health before randomization
* Has body Mass Index (BMI) between 18 and 32 kg/m2, inclusive

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has history of cancer (malignancy)
* Has positive test(s) for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in QT Interval Corrected for Heart Rate (QTc) Following Ulonivirine Administration | Baseline and up to approximately 24 hours
  Change from baseline in QTc following ulonivirine administration will be reported.
Plasma Concentration of Ulonivirine at QTc Intervals (Cqtc) | At designated timepoints (up to approximately 24 hours)
  Blood samples will be collected to determine the Cqtc of ulonivirine.

SECONDARY OUTCOMES:
Change From Baseline in QT Interval Corrected for Heart Rate (QTc) Following Moxifloxacin Administration | Baseline to up to approximately 24 hours
  Change from baseline in QTc following moxifloxacin administration will be reported.
Plasma concentration of Moxifloxacin at QTc intervals (Cqtc) | At designated timepoints (up to approximately 24 hours)
  Blood samples will be collected to determine the Cqtc of moxifloxacin.
Maximum Plasma Concentration (Cmax) of Moxifloxacin | At designated timepoints (up to approximately 168 hours)
  Blood samples will be collected to determine the Cmax of moxifloxacin.
Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) of Ulonivirine | At designated timepoints (up to 168 hours)
  Blood samples will be collected to determine the AUC0-24 of ulonivirine.
Maximum Plasma Concentration (Cmax) of Ulonivirine | At designated timepoints (up to 168 hours)
  Blood samples will be collected to determine the Cmax of ulonivirine.
Time to Maximum Plasma Concentration (Tmax) of Ulonivirine | At designated timepoints (up to 168 hours)
  Blood samples will be collected to determine the Tmax of ulonivirine.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- ICON Early Phase Services (0001), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com